CLINICAL TRIAL: NCT00330148
Title: Clinical Trial Comparing the Therapeutic Combinations Melarsoprol-Nifurtimox, Melarsoprol-Eflornithine and Eflornithine-Nifurtimox in the Treatment of Gambiense Human African Trypanosomiasis in the Meningo-Encephalitic Phase
Brief Title: Randomized Clinical Trial of Three Drug Combinations for Late-Stage Gambiense Human African Trypanosomiasis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Médecins Sans Frontières, France (Other); Embassy of France in Uganda (Unknown); National Sleeping Sickness Control Program, Uganda (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPICENTRE-BTT
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2006-05

CONDITIONS: Trypanosomiasis, African
Keywords: trypanosomiasis; gambiense; combination drug therapy; sleeping sickness; Uganda
MeSH Terms: conditions — Trypanosomiasis, African; Trypanosomiasis | interventions — Melarsoprol; Nifurtimox; Eflornithine

INTERVENTIONS:
Drug: melarsoprol 1.8 mg/kg/d, 10d + nifurtimox 15/20 mg/kg/d, 10d
Drug: melarsoprol 1.8 mg/kg/d, 10d + eflornithine 400 mg/kg/d, 7d
Drug: nifurtimox 15/20 mg/kg/d 10d + eflornithine 400 mg/kg/d 7d

SUMMARY:
The treatment human African trypanosomiasis (HAT) in the meningoencephalitic phase relies on two molecules officially registered: melarsoprol, the most commonly used, has a poor safety profile and is becoming ineffective due to parasite resistance; and eflornithine, with better tolerance but more complicated and expensive to implement in endemic countries. nifurtimox, registered only for Chagas' disease but used off-label since the 1970's in series of cases of HAT, is at present the only other available alternative.

The very limited number of compounds available, the lack of prospects for the development of new products and the emergence of resistance are arguments for the use of therapeutic combinations.

This study evaluates the efficacy and safety of three drug combination therapies: melarsoprol-nifurtimox, melarsoprol-eflornithine and eflornithine-nifurtimox.

DETAILED DESCRIPTION:
Dosages per drug are the same in either arm of the study: IV melarsoprol 1.8 mg/kg/day, daily for 10 days; IV eflornithine 400 mg/kg/day, 6-hourly for 7 days; oral nifurtimox 15 or 20 (children <15 years) mg/kg/day, 8-hourly for 10 days.

For efficacy assessment, patients are followed-up for 24 months after treatment, with planned clinical and laboratory controls.

The safety assessment includes clinical and hematological adverse events.

ELIGIBILITY:
Inclusion Criteria:

* confirmed second-stage T.b. gambiense infection :

  * Infection diagnosed parasitologically (blood or lymph node fluid) and white blood cells > 5/mm3 in cerebrospinal fluid (CSF)
  * or Trypanosomes detected in the CSF with any CSF cell count
* and resident in the district
* and written consent of the patient or of one of the parents/guardians for children under 15 years of age.

Exclusion Criteria:

* Trypanosome absent from blood (or lymph node fluid) and from CSF
* Or women pregnant on inclusion
* Or previous history of HAT confirmed treated during the last 24 months
* Or impossibility of regular access to the treatment centre during the 2 years following the end of the treatment
* Or less than 10 kg of body weight
* Or refugee patient

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 435
Dates: Start 2001-03; Study Completion 2004-06

PRIMARY OUTCOMES:
Cure rate

SECONDARY OUTCOMES:
Adverse events temporally associated with the treatment
Major adverse events temporally associated with the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Priotto, MD, MPH, Principal Investigator — Epicentre
Locations (1):
- Omugo Sleeping Sickness Treatment Center, Omugo, Arua District, Uganda

REFERENCES:
- [Background] Legros D, Ollivier G, Gastellu-Etchegorry M, Paquet C, Burri C, Jannin J, Buscher P. Treatment of human African trypanosomiasis--present situation and needs for research and development. Lancet Infect Dis. 2002 Jul;2(7):437-40. doi: 10.1016/s1473-3099(02)00321-3. PMID 12127356